CLINICAL TRIAL: NCT05329974
Title: Computer Guided Buccal Cortical Plate Separation for Removal of Calcified Benign Odontogenic Tumors Affecting Mandibular Angle Region
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Sherif Ali, Associate Professor, Cairo University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OMFS-11021
Record Dates: First submitted 2022-04-06; First posted 2022-04-15 (Actual); Last update posted 2022-04-15 (Actual); Status verified 2022-04

CONDITIONS: Odontogenic Tumors; Odontoma
MeSH Terms: conditions — Odontogenic Tumors; Odontoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Computer guided buccal cortical plate separation (Experimental): Computer guided buccal cortical plate separation for removal of calcified benign odontogenic tumors
  Interventions: Other: Computer guided buccal cortical plate separation

INTERVENTIONS:
Other: Computer guided buccal cortical plate separation — Computer guided buccal cortical plate separation for removal of calcified benign odontogenic tumors

SUMMARY:
Computer guided buccal cortical plate separation was performed for ten patients using patient specific osteotomy locating guides and pre-bent plates. The guide was designed to outline the osteotomy, buccal cortical plate was separated, the lesion was removed, finally the pre-bent plates were used to fix the separated cortex.

DETAILED DESCRIPTION:
Computer guided buccal cortical plate separation was performed for ten patients using patient specific osteotomy locating guides and pre-bent plates. The guide was designed to outline the osteotomy, buccal cortical plate was separated, the lesion was removed, finally the pre-bent plates were used to fix the separated cortex.

ELIGIBILITY:
Inclusion Criteria:

* Patients with well-defined radiopaque lesion affecting angle region, its conventional removal may compromise the bone continuity and leads to pathological fracture indicating the need of buccal cortical plate separation technique

Exclusion Criteria:

* Patients with any medical condition contraindicating the surgical procedures were excluded

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2021-07-30 (Actual); Study Completion 2021-07-30 (Actual)

PRIMARY OUTCOMES:
Intra-operative time | during the surgery
  Intra-operative time was measured from the start of the incision till suturing

SECONDARY OUTCOMES:
Postoperative pain | 2, 5, and 10 days after the surgery
  Postoperative pain using 0 - 10 visual analog scale
Edema | 5 and 10 days after the surgery
  Edema was assessed using a four grades scale: Grade 0, No edema; Grade 1, mild edema (just visible); Grade 2; moderate edema (local); Grade 3, severe edema (extended).

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - Faculty of dentistry, Cairo university, Cairo
  - Faculty of Dentistry, Cairo

REFERENCES:
- [Derived] Omara M, Gouda A, Ali S. Computer-guided buccal cortical plate separation for removal of calcified benign odontogenic tumors affecting the mandibular angle region. Maxillofac Plast Reconstr Surg. 2022 Sep 22;44(1):30. doi: 10.1186/s40902-022-00354-6. PMID 36136180